CLINICAL TRIAL: NCT03933670
Title: A Phase 2 Study of Magnetic Resonance (MR) Imaging with Hyperpolarized Pyruvate (13C) in Patients with Prostate Cancer on Active Surveillance
Brief Title: Hyperpolarized Pyruvate (13C) MR Imaging in Monitoring Patients with Prostate Cancer on Active Surveillance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Ivan de Kouchkovsky, MD, Assistant Clinical Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 175516; NCI-2018-02195 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA211150 (NIH); R01EB017449 (NIH); U01CA232320-01A1 (NIH)
Record Dates: First submitted 2019-02-20; First posted 2019-05-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Prostate Adenocarcinoma; Prostate Cancer
Keywords: Imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; Hydrogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (HP C-13 MRI) (Experimental): Patients receive hyperpolarized carbon C 13 pyruvate IV over less than one minute, then undergo MRSI after 1-2 minutes. Within 15-60 minutes, patients may receive optional hyperpolarized carbon C 13 pyruvate and undergo MRSI. Patients also undergo MR/US fusion-guided prostate biopsy within 12 weeks following HP C-13 MRSI.
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Spectroscopic Imaging; Procedure: MRI Ultrasound Fusion Guided Biopsy

INTERVENTIONS:
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: Hydrogen-1 (1H)- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging
Procedure: MRI Ultrasound Fusion Guided Biopsy — Undergo MR/US fusion-guided prostate biopsy
  Other Names: Fusion Biopsy; Fusion Guided Biopsy; Fusion-Guided Biopsy; MR Fusion Biopsy; MRI-Ultrasound Fusion Biopsy; MRI/Ultrasound Fusion Biopsy; MRI/US Biopsy

SUMMARY:
This phase II trial studies the side how well hyperpolarized carbon C 13 pyruvate (HP C-13 pyruvate) magnetic resonance imaging (MRI) works in monitoring patients with prostate cancer on active surveillance who have not received treatment. Diagnostic procedures, such as MRI, may help visualize HP C-13 pyruvate uptake and breakdown in tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Optimize the imaging sequences that maximize signal-to-noise ratio (SNR) and intra-tumoral conversion of HP 13C pyruvate to lactate (kPL) and HP 13C pyruvate to glutamate (kPG) in regions of tumor versus (vs.) adjacent benign tissue as assessed by multi-parametric MRI (mpMRI) imaging characteristics. (Part 1) II. Determine the association between intra-tumoral kPL and kPG with Gleason grade determined during magnetic resonance (MR)/ultrasound (US)-guided fusion prostate biopsies obtained within 6 months following baseline HP C-13 pyruvate MR exam. (Part 2)

SECONDARY OBJECTIVES:

I. Evaluate the intra-patient variability in intra-tumoral kPL and kPG with repeated dose studies.

II. Determine the association between peak intra-tumoral kPL observed on baseline imaging with serum prostate specific antigen (PSA).

III. Compare and contrast intra-tumoral kPL and kPG with prostate imaging reporting and data system (PI-RADS) version 2 and individual mpMRI parameters including apparent diffusion coefficient (ADC) on diffusion-weighted imaging.

IV. Describe the frequency of up-grading of tumor with MR/US-guided fusion biopsy obtained following baseline HP C-13 MR exam.

V. Further characterize the safety profile of HP C-13 pyruvate injections.

EXPLORATORY OBJECTIVES:

I. Correlate peak intra-tumoral kPL with results of gene expression profiling using DECIPHER assay.

II. Correlate peak intra-tumoral kPL and kPG with DECIPHER GRID tumor ribonucleic acid (RNA) expression of relevant components of the glycolytic pathway including lactate dehydrogenase (LDH), pyruvate dehydrogenase (PDH), aconitate hydratase (aconitase), myelocytomatosis oncogene (MYC), monocarboxylate transporter 4 (MCT4) (lactate transporter).

III. For patients who undergo optional follow-up HP C-13 pyruvate/MRI 6-15 months following baseline scan, determine the mean percent change from baseline in intra-tumoral kPL and kPG and whether the change from baseline is associated change in clinical risk assessment as determined by University of California, San Francisco (UCSF)-Cancer of the Prostate Risk Assessment (CAPRA) risk score.

OUTLINE:

Patients receive hyperpolarized carbon C 13 pyruvate intravenously (IV) over less than one minute, then undergo magnetic resonance spectroscopic imaging (MRSI) after 1-2 minutes. Within 15-60 minutes, patients may receive optional hyperpolarized carbon C 13 pyruvate and undergo MRSI. Patients also undergo MR/US fusion-guided prostate biopsy within 12 weeks following HP C-13 MRSI.

After completion of study, patients will be followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* The subject has biopsy-proven adenocarcinoma of the prostate with low to intermediate risk disease by UCSF-CAPRA scoring at study entry.
* For Part 1: Patient planning to enroll or currently on active surveillance; For Part 2: Currently enrolled on active surveillance with planned fusion biopsy within 12 weeks following completion of baseline HP C-13 pyruvate/mpMRI on study.
* The subject is able and willing to comply with study procedures and provide signed and dated informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Absolute neutrophil count (ANC) >= 1000 cells/microliter (uL).
* Hemoglobin >= 9.0 gm/deciliter (dL).
* Platelets >= 75,000 cells/uL.
* Estimated creatinine clearance* >= 50 milliliter (mL)/min by the Cockcroft Gault equation.
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if =< 3 x ULN if known/suspected Gilbert's
* Aspartate aminotransferase (AST) =< 1.5 x ULN.
* Alanine aminotransferase (ALT) =< 1.5 x ULN.

Exclusion Criteria:

* Patients without evidence of any prostate cancer on most recent prostate biopsy performed prior to study entry.
* Current or prior androgen deprivation therapy including luteinizing hormone-releasing hormone (LHRH) analogue or oral anti-androgen therapy. Previous use of a 5-alpha reductase inhibitor is allowed, provided it was discontinued at least 28 days prior to baseline C-13 HP pyruvate MRI
* Prior radiation treatment of the prostate.
* Prostate biopsy performed within 14 days prior to baseline C-13 HP pyruvate MRI.
* Poorly controlled hypertension, with blood pressure at study entry > 160 mm Hg systolic or > 100 mmg Hg diastolic. Treatment with anti-hypertensives and re-screening is permitted.
* Congestive heart failure with New York Heart Association (NYHA) status >= 2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Signal-to-noise ratio (SNR) of hyperpolarized lactate | At Baseline
  Assessed by multi-parametric magnetic resonance imaging (mpMRI) characteristics.
Intra-tumoral C-pyruvate to lactate (kPL) | At Baseline
  Assessed by multi-parametric magnetic resonance imaging (mpMRI) characteristics
Intra-tumoral C-pyruvate to glutamate (kPG) | At Baseline
  Assessed by multi-parametric magnetic resonance imaging (mpMRI) characteristics
Association between intra-tumoral C-pyruvate to lactate (kPL) with Gleason grade | Within 12 weeks following baseline HP C-13 pyruvate MR exam
  kPL will be compared with the pathologic Gleason grade determined using tissue from an MR/US-guided fusion prostate biopsy. Measured kPL will be compared by pathologic Gleason grade using an ANOVA model. If there is an overall difference, the Newman-Keuls post hoc test will be used to determine which tissue pairs differ.
Association between intra-tumoral C-pyruvate to glutamate (kPG) with Gleason grade | Within 12 weeks following baseline HP C-13 pyruvate MR exam
  kPG will be compared with the pathologic Gleason grade determined using tissue from an MR/US-guided fusion prostate biopsy. Measured kPG will be compared by pathologic Gleason grade using an ANOVA model. If there is an overall difference, the Newman-Keuls post hoc test will be used to determine which tissue pairs differ.

SECONDARY OUTCOMES:
Intra-patient variability in kPL | Up to 15 months
  Intra-patient variability in the kPL will be summarized by the intraclass correlation and presented with a 90% confidence interval.
Intra-patient variability in kPG | Up to 15 months
  Intra-patient variability in the kPG will be summarized by the intraclass correlation and presented with a 90% confidence interval.
Contrast between kPL and kPG in regions of tumor | Up to 15 months
  The kPL and kPG will be contrasted in regions of tumor. Determined with prostate imaging reporting and data system (PI-RADS) version 2 classification score (1 through 5)
Comparison of kPL and kPG with apparent diffusion coefficient in region of tumor | Up to 15 months
  The kPL and kPG will be compared with apparent diffusion coefficient in region of tumor. Determined by comparison to peak intra-tumoral apparent diffusion coefficient (ADC) value
Incidence of adverse events graded | Up to 15 months
  According to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Association between peak intra-tumoral kPL observed on baseline imaging with serum PSA | At Baseline
  Determine the association between peak intra-tumoral kPL observed on baseline imaging with serum PSA. The study cohort will be dichotomized by mean intra-tumoral kPL above and below the median and the mean serum PSA will be compared between the two dichotomized subgroups using Mann-Whitney test.
Describe frequency of up-grading of tumor | Within 12 weeks following baseline HP C-13 pyruvate MR exam
  Describe the frequency of up-grading of tumor with MR/US-guided fusion biopsy obtained following baseline HP C-13 MR exam

CONTACTS AND LOCATIONS:
Overall Officials: Ivan de Kouchkovsky, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No